CLINICAL TRIAL: NCT04574284
Title: A Open-label, Multicenter Phase II Study of TQB2450 Injection or Combined With Anlotinib Hydrochloride Capsule in Subjects With Advanced Endometrial Cancer
Brief Title: A Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule in Subjects With Advanced Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-08
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Advanced Endometrial Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2450 + Anlotinib (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450; Drug: Anlotinib
- TQB2450 (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle.
  Interventions: Drug: TQB2450
- Anlotinib (Experimental): Anlotinib capsules 12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
  Arms: TQB2450; TQB2450 + Anlotinib
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor.
  Arms: Anlotinib; TQB2450 + Anlotinib

SUMMARY:
This is a study to evaluate the efficacy and safety of TQB2450 injection or combined with anlotinib hydrochloride capsule in the treatment of recurrent or metastatic advanced endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and signed an informed consent form. 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

  3. Histopathologically confirmed recurrent or metastatic advanced endometrial cancer.

  4. Has at least one measurable lesion. 5. Agree to provide tumor tissue samples for MSI/MMR status detection. 6. Adequate laboratory indicators. 7. Serum or urine pregnancy tests are negative within 7 days before randomization; Men and women should agree to use effective contraception during the study period and after the end of the study period within 6 months.

Exclusion Criteria:

* 1.Concomitant disease and medical history:

  1. Has diagnosed and/or treated additional malignancy within 3 years prior to randomization;
  2. Pathological diagnosed as uterine sarcoma;
  3. Has multiple factors affecting oral medication;
  4. Unalleviated toxicity ≥ grade 1 due to any previous anticancer therapy.
  5. Has received major surgical treatment, open biopsy and so on within 28 days before the start of the study.
  6. Has a unhealed wound or fracture for a long time;
  7. Has cerebrovascular accident, deep vein thrombosis and pulmonary embolism within 6 months before the study;
  8. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures;
  9. Has a history of psychotropic substance abuse and unable to quit or mental disorders;
  10. Has any serious and / or uncontrolled disease; 2. Tumor-related symptoms and treatment:

  <!-- -->

  1. Has received surgery, chemotherapy, radiotherapy or other anticancer therapy within 4 weeks before the start of the study;
  2. Has received proprietary Chinese medicine with anti-tumor indications in the NMPA approved drug instructions within 2 weeks before the start of the study;
  3. Has received immunotherapeutic drugs against PD-1, PD-L1, CTLA-4 and other related drugs;
  4. Has used antiangiogenic drugs such as bevacizumab, anlotinib, apatinib, lenvatinib, sorafenib, Sunitinib, regorafenib, fruquintinib, etc;
  5. Has received hormone therapy for endometrial cancer within a week before the first dose ;
  6. CT or MRI showed that the tumor had invaded the important blood vessels;
  7. Has symptomatic central nervous system (CNS) disease and/or cancerous meningitis, pia mater disease; 3. Related to research and treatment:

  <!-- -->

  1. Has received attenuated live vaccine within 28 days before randomization or planned to received attenuated live vaccine during the study period.
  2. Has a history of severe allergic diseases.
  3. Has active autoimmune diseases requiring systemic treatment occurred within 2 years before the study.

     4. Has Participated in other clinical trials within 4 weeks before first dose. 5. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) evaluated by Independent Review Committee(IRC) | up to 12 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR), recorded from the first dose until the first documented progressive disease (PD) or death from any cause, based on IRC.

SECONDARY OUTCOMES:
Overall response rate (ORR) evaluated by investigator | up to 12 months
  ORR defined as percentage of participants achieving complete response (CR) and partial response (PR), recorded from the first dose until the first documented progressive disease (PD) or death from any cause, based on investigator.
Disease control rate (DCR) | up to 12 months
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of response (DOR) | up to 12 months
  The time when the participants first achieved complete or partial remission to disease progression.
Progression free survival(PFS) | up to 12 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Overall survival(OS) | up to 18 months
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
DOR rate (≥ 6 months) | up to 6 months
  The percentage of participants achieved complete or partial remission ≥ 6 months.

CONTACTS AND LOCATIONS:
Locations (36):
- China (36):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tsinghua University Affiliated Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Gansu Province Maternity and Chid-care Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an People's Hospital, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital, School of Medicine, Shihezi University, Shihezi, Xinjiang Uygur Autonomous Region
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang Uygur Autonomous Region
  - Xinjiang Medical University Affiliated Tumor Hospital, Ürümqi, Xinjiang Uygur Autonomous Region
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang